CLINICAL TRIAL: NCT01659788
Title: Co Enzyme Q10 Improves IVF Outcome in With Advanced Reproductive Age
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CoEnzyme Q10-HMO-CTIL
Record Dates: First submitted 2012-08-05; First posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Ovarian Function at Advanced Reproductive Age
Keywords: Advanced Reproductive Age; poor ovarian response; Mitochondrial dysfunction; Mitochondrial nutrients; Coenzyme Q10; Electron transfer chain
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coenzyme Q10 concomitant treatment (Experimental): Coenzyme Q10 concomitant treatment to fertility drugs as part of an IVF treatment
  Dose: 600 mg by mouth daily beginning 3 months prior to IVF cycle. Patient will stop taking the CoEnzyme Q10 if conceives or when the study is completed.
  Other name: Ubiquinone
  Interventions: Dietary Supplement: Coenzyme Q10 concomitant treatment
- Placebo (Placebo Comparator): 1 capsule by mouth daily beginning 3 months prior to IVF cycle. Patient will stop taking the placebo when she conceives or when the study is completed.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 concomitant treatment
  Arms: Coenzyme Q10 concomitant treatment
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The goal of the investigators research is to explore energy production of the ovarian follicle in older reproductive age women at the time of oocyte retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Age 38-43 years at the time of enrollment
* Diagnosis of primary infertility

Exclusion Criteria:

* Body mass index (BMI) > 30 kg/m2
* Early follicular phase (day 2-4) serum FSH level > 20 mIU/ml.
* Abnormal uterine cavity as evidenced by sonohysterogram or hysterosalpingography
* Any current use of systemic steroid medication or any infertility treatment within 3 months of study enrollment.
* Any contraindication to being pregnant and carrying a pregnancy to term.
* Contraindication for the use of CoQ10, or fertility medications.
* Any ovarian or abdominal abnormality that may interfere with adequate TVS evaluation.
* Absence of one or two ovaries
* Clinically relevant systemic disease (e.g., Insulin-dependent diabetes, adrenal dysfunction, organic intracranial lesion, polycystic ovarian syndrome, hyperprolactinemia, or hypothalamic tumor) or serious illness (Neoplasia).
* History (within past 12 months) or current abuse of alcohol or drugs.
* Administration of any investigational drugs within three months prior to study enrollment.
* Any medical condition that may interfere with the absorption, distribution, metabolism or excretion of the study drugs, gastrointestinal diseases, mal absorption syndromes and liver dysfunction
* Unexplained gynecological bleeding.
* Ejaculated sperm is not sufficient for ICSI
* Patient not able to communicate adequately with the investigators and to comply with the requirements of the entire study.
* Abnormal COH screening blood done for both partners, including: prolactin, thyroid stimulating hormone, HIV serology, Hepatitis B and C serology, Rubella, group and screen and syphilis serology prior to participation in study.
* Unwillingness to give written informed consent. Previous entry into this study or simultaneous participation in another clinical trial.
* The concurrent use of any of the following drugs:
* Daunorubicin, Doxorubicin, Blood Pressure Medications, Warfarin, Timolol, atorvastatin, cerivastatin, lovastatin, pravastatin, simvastatin gemfibrozil, tricyclic antidepressant medications (including amitriptyline, amoxapine, clomipramine, desipramine, doxepin, imipramine, nortriptyline, protriptyline, and trimipramine) multivitamins or any vitamin supplementation except Folic acid.

Ages: 38 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
level of ATP production | 2 years
Steriodogenesis associated enzymatic activity | 2 years

SECONDARY OUTCOMES:
Ovarian Response | 2 years
Embryo quality | 2 years
cumulative pregnancy rate per retrieval | 2 years
cumulative live birth rate per retrieval | 2 years

OTHER OUTCOMES:
Co Enzyme Q10 levels in maternal serum by HPLC | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Kochman, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel